CLINICAL TRIAL: NCT02247674
Title: Effects of Computer-aided Interlimb Force Coupling Training on Paretic Hand and Arm Motor Control Following Chronic Stroke
Brief Title: Bilateral Movement Training for People With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chueh-Ho Lin (Other)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor-Investigator, Chueh-Ho Lin, Dr., National Yang Ming Chiao Tung University
Organization: National Yang Ming Chiao Tung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYMU20140829
Record Dates: First submitted 2014-08-31; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Stroke; Cerebrovascular Accident; Cardiovascular Disease; Brain Injury
Keywords: Stroke, Cerebrovascular accident, Rehabilitation, Upper extremity
MeSH Terms: conditions — Stroke; Cardiovascular Diseases; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education & training consultation (Placebo Comparator): Education and training consultations were provided for subjects in control group during study period.
  Interventions: Procedure: Bilateral movement training
- Bilateral movement training (Experimental): Exercise training of bilateral isometric handgrip force training group consisted of 60 minutes of bilateral isometric handgrip force training 3 days per week for 4 weeks (total 12 sessions)
  Interventions: Procedure: Bilateral movement training

INTERVENTIONS:
Procedure: Bilateral movement training — Exercise training of bilateral isometric handgrip force training group consisted of 60 minutes of bilateral isometric handgrip force training 3 days per week for 4 weeks (total 12 sessions)
  Other Names: Coupling movement

SUMMARY:
The investigators hypothesized that bilateral handgrip force training would result in significant improvements in paretic hand, arm movements and daily functional performances. In order to investigate whether the improvement of paretic hand could facilitate the motor recovery of paretic arm and functional performances, the investigators also hypothesized that motor recovery and functional performances improvements of paretic arm and hand have strongly correlation.

DETAILED DESCRIPTION:
Objective: To investigate the training effects of interlimb force coupling training on paretic hand and upper extremity outcomes in patients with chronic stroke; to analyze the relationship between motor recovery of paretic hand, arm and functional abilities.

Design: A double-blind randomized controlled trial with outcome assessment at baseline and after 4 weeks intervention.

Setting: Department of physical medicine and rehabilitation in Taipei Veterans General Hospital.

Participants: Thirty-three subjects (mean age = 55.1 ± 10.5 y/o) with chronic stroke were recruited and randomized assigned to training (n=16) and control group (n=17).

Interventions: Interlimb force coupling training task included different gripforce generation on the both hands.

Main Outcome Measures: Barthel Index (BI), and the upper extremity motor control of Fugl-Meyer Assessment (FMA-UE), Motor Assessment Score (MAS), and the Wolf Motor Function Test (WMFT). All assessment was executed by a blinded evaluator, and data management and statistical analysis was also conducted by a blinded statistic researcher.

ELIGIBILITY:
Inclusion Criteria:

1. at least 6 months since stroke
2. three or fewer incidents of unilateral stroke confirmed by taking the participant's medical history ability to follow researcher's instructions
3. ability to flex and extend the paretic arm and hand
4. Modified Ashworth Score (MAS) ≦3 for wrist and finger joints
5. Mini-Mental State Examination (MMSE) score should 24 or higher
6. no other orthopedic neurological disorders
7. Brunnstrom stage 3 or 4
8. no joint in other experimental rehabilitation or drug studies 21

Exclusion Criteria:

1. unstable cardiovascular conditions
2. uncontrolled hypertension (190/110 mm Hg)
3. severe orthopedic or pain conditions
4. dementia (Mini-Mental State Examination score < 22)
5. aphasia with inability to follow researcher's commands
6. severe joint contracture of bilateral upper extremities that would impact the movement performances of upper extremities

Ages: 28 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Upper Extremity motor control of Fugl-Meyer Assessment (FMA-UE) | before and after 4 weeks intervention
  Outcome measure was assessed before and after 4 weeks intervention.

SECONDARY OUTCOMES:
Barthel Index (BI) | before and after 4 weeks intervention
  Outcome measure was assessed before and after 4 weeks intervention.
Motor Assessment Score (MAS) | before and after 4 weeks intervention
  Outcome measure was assessed before and after 4 weeks intervention.
Wolf Motor Function Test (WMFT) | before and after 4 weeks intervention
  Outcome measure was assessed before and after 4 weeks intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hsu Sung, PhD, Study Chair — Department of Physical Therapy and Assistive Technology, National Yang-Ming University
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin CH, Chou LW, Luo HJ, Tsai PY, Lieu FK, Chiang SL, Sung WH. Effects of Computer-Aided Interlimb Force Coupling Training on Paretic Hand and Arm Motor Control following Chronic Stroke: A Randomized Controlled Trial. PLoS One. 2015 Jul 20;10(7):e0131048. doi: 10.1371/journal.pone.0131048. eCollection 2015. PMID 26193492